CLINICAL TRIAL: NCT07050563
Title: Clinical Evaluation of the Tiaoshen Anti-Cancer Regimen in Treating Psycho-Neurological Symptom Cluster in Ovarian Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Affiliated Hospital of Qinghai University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Fudan University (Other); Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024ZD0521402
Record Dates: First submitted 2025-06-11; First posted 2025-07-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Cancer Symptom Clusters
MeSH Terms: conditions — Neoplasms | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Daily Compound Ciwujia granules+ standard treatment protocol for ovarian cancer+ psychological intervention
  Interventions: Drug: Compound Ciwujia Granules; Combination Product: Standard treatment protocol for ovarian cancer combined with psychological intervention.
- Control group (Placebo Comparator): Daily placebo granules + standard treatment protocol for ovarian cancer+ psychological intervention
  Interventions: Drug: Placebo granules; Combination Product: Standard treatment protocol for ovarian cancer combined with psychological intervention.

INTERVENTIONS:
Drug: Compound Ciwujia Granules — In addition to standard treatment protocol for ovarian cancer combined with psychological intervention, Compound Ciwujia Granules were administered at a dosage of one sachet twice daily for a treatment duration of 3 months.
  Arms: Intervention Group
Drug: Placebo granules — In addition to standard treatment protocol for ovarian cancer combined with psychological intervention, placebo granules which containing 10% of Compound Ciwujia Granules drug were administered at a dosage of one sachet twice daily for a treatment duration of 3 months.
  Arms: Control group
Combination Product: Standard treatment protocol for ovarian cancer combined with psychological intervention. — Standard treatment protocol for ovarian cancer: In accordance with the 2024 NCCN International Guidelines, patients opt for chemotherapy regimens containing platinum-based drugs and/or targeted therapy, anti-angiogenic therapy, hormonal therapy, etc. Psychological intervention is conducted once a week in the form of online and offline patient education sessions for psychological intervention, continuing until the end of the study period. Both the intervention group and the control group use this as the baseline treatment plan.

SUMMARY:
The academic community generally believes that cancer symptom clusters (CSCs) are not independent diseases, but a group of symptoms that accompany cancer patients. Based on etiology, they can be classified into CSCs related to tumor progression, CSCs related to cancer treatment, or a combination of both. According to symptom manifestations, they can be divided into psychological symptom CSCs, somatic symptom CSCs, and CSCs with coexisting psychological and somatic symptoms. CSCs are universally present during the progression or treatment of cancer. Traditional Chinese medicine (TCM) can leverage its unique characteristics in the intervention of symptom clusters and symptom management. This study is planned to conduct a high-level, prospective, multicenter, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of a TCM regimen for cancer symptom clusters (CSCs), and to simultaneously analyze the characteristics of the population that may benefit most from TCM treatment for CSCs.

DETAILED DESCRIPTION:
Targeting ovarian cancer patients with psychoneurological symptom clusters, a multicenter, randomized, placebo-controlled, superiority clinical trial was conducted. On the basis of psychological intervention and conventional cancer treatment, the treatment group and the control group respectively received Compound Ciwujia Granules or a placebo. The intervention lasted for three months, with the alleviation of psychoneurological symptoms assessed before and after treatment in both groups.

The primary efficacy endpoint was the mean score of the subscale comprising sleep disturbance, fatigue, distress, and sadness from the Chinese version of the MD Anderson Symptom Inventory for Ovarian Cancer (MDASI-OC). Secondary efficacy endpoints included the EORTC QLQ-C30 quality of life scale, sleep quality assessment, and sleep diaries. Exploratory endpoints included the 1-year overall survival (OS) rate and progression-free survival (PFS) rate. Peripheral blood samples and tumor tissue specimens were collected to investigate common biological targets underlying the psychoneurological symptom cluster in ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary epithelial ovarian cancer
* Meet diagnostic criteria for chronic insomnia defined by the Sleep Disorders Group of the Neurology Branch of the Chinese Medical Association: Pittsburgh Sleep Quality Index (PSQI) total score >8 Piper Fatigue Scale total score >4 and Patient Health Questionnaire-9 (PHQ-9) total score >5
* Moderate-to-severe symptom severity (average score ≥4 on the MD Anderson Symptom Inventory for Ovarian Cancer [MDASI-OC] subscale assessing sleep disturbance-fatigue-distress-sadness)
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score 0-2;
* Age 18-70 years
* Meeting TCM diagnostic criteria for spleen-kidney yang deficiency syndrome;
* Expected survival >1 year
* Signed informed consent form with voluntary acceptance of the treatment protocol and ability to independently complete sleep diaries

Exclusion Criteria:

* Patients scheduled to undergo radiotherapy within the next 4 treatment cycles
* Comorbid severe primary diseases of the heart, brain, liver, kidney, or hematopoietic system, including hepatic dysfunction (AST/ALT >1.5 times the upper limit of normal [ULN]) or renal impairment (serum creatinine [Cr] >1.2 times ULN)
* Pregnant or lactating women, individuals with psychiatric disorders (e.g., schizophrenia, bipolar disorder, mania, depression, anxiety disorders, phobias), intellectual/language impairments, or other mental health conditions;
* Scores ≥15 on the Patient Health Questionnaire (PHQ-9) for depression or ≥15 on the Generalized Anxiety Disorder-7 (GAD-7) at screening
* Pre-existing chronic insomnia or depression diagnosed prior to ovarian cancer
* Comorbid autoimmune diseases, hematologic disorders, or long-term use of corticosteroids/immunosuppressants
* History of other primary malignancies
* Participation in other clinical trials within 3 months
* HIV-positive status, congenital/acquired immunodeficiency disorders, or history of organ transplantation (including autologous bone marrow or peripheral stem cell transplantation)
* Legally incapacitated individuals, or cases with medical/ethical contraindications to study continuation
* Active hepatitis B, active tuberculosis, or evidence of severe/uncontrolled systemic inflammatory conditions (e.g., unstable respiratory, cardiovascular, hepatic, or renal diseases)
* Patients with diabetes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Psychoneurological Symptom Cluster in Ovarian Cancer | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  Mean score of the subscale composed of sleep disturbance, fatigue, distress, and sadness in the MD Anderson Symptom Inventory for ovarian cancer (MDASI-OC)

SECONDARY OUTCOMES:
Piper Fatigue Scale | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
Pittsburgh Sleep Quality Index (PSQI) Sleep Scale | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
Patient Health Questionnaire-9 (PHQ-9) Depression Scale | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
Chinese Traditional Medicine Syndrome Pattern Assessment Scale | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
EORTC QOL-C30 Scale | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  Quality of Life Questionnaire-Core 30
Generalized Anxiety Disorder 7-item (GAD-7) Anxiety Scale | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  It is a self-assessment tool used to evaluate the severity of anxiety symptoms, consisting of 7 questions with a total score ranging from 0 to 21 points. It can be divided into 4 grades, and the higher the score, the more severe the condition
1-year survival analysis | Determined at the 1-year follow-up after random assignment
  From randomization, patients underwent regular imaging assessments to determine 1-year overall survival (OS) and progression-free survival (PFS) rates.

OTHER OUTCOMES:
Sleep quality | Assessments at baseline and at 1, 2, and 3 months post-enrollment
  Assessing sleep quality using a portable wristband.
Sleep diary | Assessments at baseline and at 1, 2, and 3 months post-enrollment
  Record basic sleep metrics, such as daily bedtime, sleep onset time, number and duration of nighttime awakenings, and morning wake-up time.
Functional magnetic resonance imaging (fMRI) | Assessed at baseline and 3 months post-enrollment
  Functional magnetic resonance imaging (fMRI) is planned for 30 randomly selected patients per group, totaling 60 participants.
Biological targets in peripheral blood | Assessments at baseline and 3 months post-enrollment
  Using targeted proteomics, we detect differential protein expression in cancer patients with psychoneurological symptom clusters before and after treatment, with the goal of exploring potential actionable therapeutic targets. The study is to randomly select 50 cases from each group, totaling 100 patients for examination.
Biological targets in tumor tissue | Tumor tissue is collected exclusively at baseline
  Utilizing exclusively pre-treatment tumor tissues, we performed targeted proteomics to detect differential protein expression between cancer patients exhibiting psychoneurological symptom clusters and cancer-free healthy controls. The study plan to randomly select 50 cases from each group, totaling 100 patients for examination.
Heart rate | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  Safety indicator
Respiration | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  Safety indicator
Body temperature | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  Safety indicator
Blood pressure | Assessments at baseline and at 1, 2, 3, 6, 9 and 12 months post-enrollment
  Safety indicator
Alanine Aminotransferase (ALT) | At baseline and 3 months after enrollment
  Safety indicator
Aspartate Aminotransferase(AST) | Assessed at baseline and 3 months post-enrollment
  Safety indicator
Serum creatinine | Assessed at baseline and 3 months post-enrollment
  Safety indicator
Urinary protein | Assessed at baseline and 3 months post-enrollment
  Safety indicator
Urinary leukocytes | Assessed at baseline and 3 months post-enrollment
  Safety indicator
White blood cells (WBC) | Assessed at baseline and 3 months post-enrollment
  Safety indicator
Hemoglobin (Hb) | Assessed at baseline and 3 months post-enrollment
  Safety indicator
Platelets (PLT) | Assessed at baseline and 3 months post-enrollment
  Safety indicator
Adrenocorticotropic hormone (ACTH) | Assessed at baseline and 3 months post-enrollment
  As indicator for assessing Hypothalamic-Pituitary-Adrenal(HPA) axis function, assayed via blood sampling.
  The study is to randomly select 50 cases from each group, totaling 100 patients for examination
Urinary free cortisol | Assessed at baseline and 3 months post-enrollment
  As indicator for assessing Hypothalamic-Pituitary-Adrenal(HPA) axis function, assayed via urine sampling.
  The study is to randomly select 50 cases from each group, totaling 100 patients for examination
Plasma cortisol | Assessed at baseline and 3 months post-enrollment
  As indicators for assessing Hypothalamic-Pituitary-Adrenal(HPA) axis function, assayed via blood sampling.
  The study is to randomly select 50 cases from each group, totaling 100 patients for examination.
Proportions of immune cells | Assessed at baseline and 3 months post-enrollment
  Measure the proportions of immune cells such as T cells, B cells, and natural killer (NK) cells. The study is to randomly select 50 cases from each group, totaling 100 patients for examination.
Cytokine levels | Assessed at baseline and 3 months post-enrollment
  Measure the expression levels of cytokines such as IL-6, IL-10, TNF-α, and IFN-γ. The study is to randomly select 50 cases from each group, totaling 100 patients for examination.
Immune gene expression analysis | Assessed at baseline and 3 months post-enrollment
  Perform RNA sequencing analysis on patient samples to investigate expression changes in immune-related genes, with a specific focus on their roles in immune regulation. The study is to randomly select 50 cases from each group, totaling 100 patients for examination.
Tumor marker CA-125 | Assessments at baseline and 3 months post-enrollment
  The unit of CA125 is U/ml. Indicators exceeding the normal range indicate a poor prognosis
Tumor marker Humanepididymisprotein4 (HE4) | Assessments at baseline and 3 months post-enrollment
  The unit of HE4 is pmol/l. Indicators exceeding the normal range indicate a poor prognosis
Electrocardiogram | Assessments at baseline and 3 months post-enrollment
  QT interval, as a safety indicator

CONTACTS AND LOCATIONS:
Overall Officials: Jianhui Tian, Doctor, Study Director — Shanghai Municipal Hospital of Traditional Chinese Medicine - Oncology Research Center

IPD SHARING:
Plan to Share IPD: Undecided